CLINICAL TRIAL: NCT04635345
Title: A Pilot Study Assessing the Feasibility of Using Clitoral Vibrators to Aid Vaginal Dilator Therapy in Women Presenting to Psychosexual Services With Vaginismus.
Brief Title: Feasibility of Use of Vibrators With Vaginal Dilators for Vaginismus. (Vibrator Therapy and Dilators in Vaginismus)
Acronym: ViTaDiVa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 278027
Record Dates: First submitted 2020-08-03; First posted 2020-11-19 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Vaginismus
MeSH Terms: conditions — Vaginismus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibrator Therapy + dilator/standard therapy (Experimental): Patient will receive standard therapy (initial appointment, referral for womens health physiotherapy or psychosexual counselling as standard, together with vadinal dilators and lidocaine gel) plus an external vibrator.
  Interventions: Other: External Vibrator - patient-administered.; Other: Standard care
- Dilator/standard therapy (Active Comparator): Patient will receive standard therapy (initial appointment, referral for womens health physiotherapy or psychosexual counselling as standard, together with vadinal dilators and lidocaine gel).
  Interventions: Other: Standard care

INTERVENTIONS:
Other: External Vibrator - patient-administered. — Patient provided with external vibrator for self-use, as well as vaginal dilators.
  Arms: Vibrator Therapy + dilator/standard therapy
Other: Standard care — Dilators, lidocaine topical gel, referral to psychotherapy, group therapy or womens health physio if required, self-help resources.

SUMMARY:
The acceptability of vulvar vibration therapy has been evaluated in women with vulvodynia, and found to be acceptable, however has not been assessed in women with a primary complaint of vaginismus.

This proposed study looks at the feasibility and acceptability of using clitoral vibration therapy, alongside current therapy, for women with vaginismus. It is likely that many, if not most, of these women will also have an element of vulvodynia. The investigators propose that the use of external clitoral or vulval vibration therapy is likely to be acceptable in most women with vaginismus, based on acceptability of vulvar vibration therapy in women with vulvodynia.

It is proposed that vibrator therapy may help women with female sexual dysfunction to use vaginal dilators.

DETAILED DESCRIPTION:
This is a nonrandomized controlled trial, with the initial cluster of patients receiving standard therapy, and the second cluster receiving standard therapy plus vibrator. Recruitment will be an initial 15 participants who will receive standard therapy, and then another 15 who will receive an external vibrator.

This study will take place over approximately 12 months. Enrollment of patients will be from a joint psychosexual clinic led by a medical doctor and a clinical psychologist. Female patients are referred to this clinic by General Practitioners, from within the Sexual Health service, or via Gynaecologists, frequently with complaint of difficulty or pain with penetrative sex. Exclusion criteria will be: patients unable/ unwilling to consent, transgender male or on testosterone therapy, unable to understand written and/or verbal English, current dermtatological skin conditions requiring active treatment, genital herpes simplex virus within 3 months, or not reporting symptoms of vaginismus with no evidence of vaginismus on clinical examination.

Trial information will be given at the initial appointment. If the patient wishes to enrol, than an initial baseline questionnaire will be given, and a follow up questionnaire will be filled out by phone contact at 3-4 months afterward the initial consultation at the patients consent.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent (additional measures have to be in place if children, vulnerable adults or adults unable to give consent are included)
* Female
* Over the age of 18
* With symptoms and clinical signs consistent with vaginismus/ vaginismus and vulvodynia.

Exclusion Criteria:

* Unwilling or unable to give consent
* Transgender male / on testosterone therapy
* Inability to understand written and / or verbal English
* Current dermatological skin conditions requiring active treatment
* Genital herpes simplex virus symptoms within preceding 3 months
* Not reporting symptoms of vaginismus, and no evidence of vaginismus on clinical examination.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jess Gaddie, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Ambrose King Sexual Health Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vibrator Therapy + Dilator/Standard Therapy | Dilator/Standard Therapy
Started | 15 | 15
Completed | 10 | 9
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibrator Therapy + Dilator/Standard Therapy | Dilator/Standard Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 24.7 [23 to 32] | 28.7 [21 to 37] | 26.7 [21 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Is Vibration Therapy (Through the Use of Handheld External Vibrators on Clitoral and Vulval Area) Acceptable to Women as Part of Medical Management of Vaginismus and Vaginismus/Vulvodynia, Alongside Current Medical Management?
Description: A 5-point Likert scale was used. Respondents replied to statements 'Overall I found using the (dilators/vibrator) acceptable" 1=not at all 2=a little 3=neither yes or no 4=mostly 5=completely. Intervention group mean scores listed in table. A higher score indicates increased acceptability.
  Acceptability of vibrators could not be assessed in the dilator/standard therapy group, because this group did not receive vibrators.
Time Frame: Follow up was over 6-24 months following initial contact. This allowed for any therapy including group therapy to be completed. Mean from initial to follow up was 10 months for intervention group and 11.5 months for control group.
Population: 5 patients in intervention group and 6 in control group were lost to follow up.
Measure: Mean (Standard Deviation); unit: mean score
Arm/Group | Vibrator Therapy + Dilator/Standard Therapy
Number analyzed (Participants) | 10
mean score | 4.3 (0.67)

2. Secondary Outcome: Does the Use of Clitoral/ Vulval Vibrators Help Women to Progress More Easily With the Use of Vaginal Dilators Compared to Women Not Using These?
Description: Respondents were asked to respond to statements with another 5-point Likert scale. 1=Not at all 2=not really 3=yes to some extent 4=agree 5=strongly agree. A higher score indicates a more positive outcome. In response to the statement 'the dilators have helped me manage my symptoms' those who 'agreed to some extent', 'agreed' or 'strongly agreed', numbers are listed in table.
Time Frame: as for outcome 1
Population: 15 in each group; 11 were Lost to Follow up in total
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrator Therapy + Dilator/Standard Therapy | Dilator/Standard Therapy
Number analyzed (Participants) | 10 | 9
Participants | 6 | 7

3. Secondary Outcome: Is There Any Self-reported Difference in Experiences of Pleasure or Enjoyment Around Sexual Experiences in the Two Groups of Women as Reported by FSDS (Female Sexual Distress Scale) Scores?
Description: The Female Sexual Distress Scale or FSDS is a 13-item questionnaire designed to measure sexually related personal distress, including the psychological impact of sexual dysfunction, and feelings of anger, frustration, worry related to sex. A higher score indicates more severe sexual dysfunction. The scale has a minimum score of 0 and maximum of 52.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vibrator Therapy + Dilator/Standard Therapy | Dilator/Standard Therapy
Number analyzed (Participants) | 10 | 9
score on a scale
  pre intervention FSDS | 31.80 (10.97) | 29.67 (5.56)
  post intervention FSDS | 25.90 (8.72) | 17.89 (7.78)

4. Secondary Outcome: Is There Any Self-reported Difference in Experiences of Pleasure or Enjoyment Around Sexual Experiences in the Two Groups of Women as Reported by FSFI (Female Sexual Function Index) Scores?
Description: A score of below 26.55 on the Female Sexual Function Index indicates Female Sexual Dysfunction. A lower score indicates greater sexual dysfunction. The minimum score is 2 and the maximum is 36. The FSFI is a 19-item questionnaire which uses 5-point Likert scales to investigate different domains of desire, arousal, lubrication, orgasm, satisfaction and pain. FSFI gives a score out of 36 with severe FSD (2-7.2), moderate (7.3-14.4), mild to moderate (14.5-21.6), mild (21.7-28.1) and no FSD (28.2-36). Each domain is weighted, resulting in an overall score of sexual function but can also be analysed separately.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vibrator Therapy + Dilator/Standard Therapy | Dilator/Standard Therapy
Number analyzed (Participants) | 10 | 9
score on a scale
  Pre-intervention score FSFI | 17.15 (7.5) | 21.53 (2.74)
  post intervention score FSFI | 20.01 (8.09) | 22.62 (7.52)

ADVERSE EVENTS:
Time Frame: 6-24 months (intervention mean 10 months, control group mean 11.5 months) From initial contact to final interview.
Description: Patents were encouraged to report adverse events via email or contact with research team through study completion, as per study duration above, no events reported.
Arm/Group | Vibrator Therapy + Dilator/Standard Therapy | Dilator/Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT04635345/Prot_000.pdf